CLINICAL TRIAL: NCT05959408
Title: Assessment of Bacterial Sexually Transmitted Infections (STIs) Viability by Polymerase Chain Reaction (PCR) in Men Who Have Sex With Men
Brief Title: Bacterial Sexually Transmitted Infections (STIs) Viability by Polymerase Chain Reaction (PCR)
Acronym: VISTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/52
Record Dates: First submitted 2023-04-14; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Men Who Have Sex With Men
Keywords: Chlamydia trachomatis; Neisseria gonorrhoeae; Mycoplasma genitalium; viability PCR; Nucleic acid amplification tests
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Intervention Model Description: It is a cross-sectional, without risk or constraint, monocentric study on the viability of the main bacterial STIs in MSM.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- men who have sex with men (Experimental)
  Interventions: Procedure: Collection of throat swab; Procedure: Collection of anal swab; Procedure: Collection of first void urine

INTERVENTIONS:
Procedure: Collection of throat swab — Introduction of a cotton swab for self-collection
Procedure: Collection of anal swab — Introduction of a cotton swab for self-collection
Procedure: Collection of first void urine — first void urine collected on urine pot

SUMMARY:
It is a cross-sectional, without risk or constraint, monocentric study on the viability of the main bacterial sexually transmitted infections (STIs) in men who have sex with men (MSM).

The main objective is to evaluate the proportion of pharyngeal, urogenital and anal specimens detected positive by nucleic acid amplification test (NAAT) for Chlamydia trachomatis, Neisseria gonorrhoeae and Mycoplasma genitalium that contain viable bacteria in MSM.

DETAILED DESCRIPTION:
Screening for C. trachomatis and N. gonorrhoeae STIs at 3 anatomical sites, i.e. pharyngeal, urogenital and anal, is recommended every three to six months in MSM with high-risk sexual behaviors, using NAAT. A positive NAAT result defines the patient as infected, and the patient will receive antibiotic treatment. However, repeated use of antibiotics has led to the emergence of multi-drug resistant strains of M. genitalium, another STI agent, and N. gonorrhoeae, and to changes in the gut microbiota. One disadvantage of NAATs is that they amplify the nucleic acids of viable and dead bacteria. Thus, it is not possible to affirm that the patient has an "active" infection, defined by the presence of viable bacteria. Bacterial viability can be studied by real-time PCR (called V-PCR). This method combines the high sensitivity and specificity of PCR with the ability to exclude detection of nucleic acid remnants from non-viable bacteria. It does so by incorporating a sample pretreatment step with a membrane impermeable DNA intercalating dye prior to molecular analysis by blocking amplification of remnant DNA from non-viable bacteria. This allows the V-PCR analysis to detect DNA originating from intact (i.e. viable) bacteria. Using V-PCR, studies in women have shown that only half of the anorectal samples and one quarter of the pharyngeal samples positive for C. trachomatis contain viable bacteria.

The team proposes to investigate the presence of viable C. trachomatis, N. gonorrhoeae and M. genitalium bacteria by V-PCR in pharyngeal, urogenital and anal specimens from MSM detected as positive by NAAT for these bacteria.

The results of this work will allow us to assess whether all types of specimens tested in these patients contain viable bacteria, and if so, in what proportions.

ELIGIBILITY:
Inclusion Criteria:

* Males > 18 years
* Men who have sex with men
* Participant consulting at the Bordeaux University Hospital
* Oral consent to participate in the study
* Member or beneficiary of a social security system

Exclusion Criteria:

* Participant < 18 years
* Participant subject to a legal protection measure (protection of the court, guardianship or curator).
* Participant deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of pharyngeal, urogenital, and anal specimens that contain viable C. trachomatis, N. gonorrhoeae, and M. genitalium bacteria detected by V-PCR out of all specimens containing these same bacteria detected by NAAT in MSM | Day 1
  The quantitative real-time PCR, performed on the aliquots, will target the bacteria detected by NAAT on the native sample. The quantitative real-time PCR will be performed on the Light Cycler 480 (Roche Diagnostics); the calibration curve will permit to quantify the bacterial load (result expressed in equivalent genomes per mL).

SECONDARY OUTCOMES:
Ratio of the number of participants testing positive by NAAT and V-PCR, respectively, for C. trachomatis, N. gonorrhoeae, and M. genitalium at at least one site to the total number of participants. | Day 1
  Prevalence of C. trachomatis, N. gonorrhoeae, and M. genitalium infections detected by NAAT versus V-PCR calculated
Ratio of the number of pharyngeal, urogenital, and anal specimens testing positive for C. trachomatis, N. gonorrhoeae, or M. genitalium by NAAT and V-PCR, respectively, to the total number of pharyngeal, urogenital, and anal samples collected | Day 1
  Prevalence of C. trachomatis, N. gonorrhoeae, and M. genitalium infections detected by NAAT versus V-PCR calculated
Evaluate the rate of participants who received antibiotic treatment in the absence of viable bacteria in the sample out of all treated participants. | Day 1
  Number of participants who will have received antibiotic treatment in the absence of viable bacteria divided by the total number of participants with a positive NAAT result.
Ratio of bacterial load of viable bacteria to total bacterial load (viable and nonviable bacteria) in each specimen. | Day 1
  Ratio of bacterial load of viable bacteria determined by quantitative real-time PCR (gEq/µL) to total bacterial load (viable and nonviable bacteria) determined by quantitative real-time PCR (gEq/µL) in each specimen.
Ratio of the number of N. gonorrhoeae resistant to penicillin G, cefixime, ceftriaxone, azithromycin, tetracycline, spectinomycin and ciprofloxacin to the number of N. gonorrhoeae strains tested. | Day 1
  Prevalence of N. gonorrhoeae resistance to penicillin G, cefixime, ceftriaxone, azithromycin, tetracycline, spectinomycin, and ciprofloxacin assessed by the ratio of the number of N. gonorrhoeae resistant to penicillin G, cefixime, ceftriaxone, azithromycin, tetracycline, spectinomycin and ciprofloxacin to the number of N. gonorrhoeae strains tested.

CONTACTS AND LOCATIONS:
Overall Officials: Charles CAZANAVE, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Olivia PEUCHANT, PharmD, Study Director — University Hospital, Bordeaux
Locations (1):
- Service des Maladies Infectieuses et Tropicales, Hôpital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No